CLINICAL TRIAL: NCT02857608
Title: A Prospective, Open-Label, Multi-center Comparison of Lymphoseek Identified Lymph Nodes and Clinically Identified Lymph Nodes of Subjects With Known Cancer of the Anus
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Cardinal Health 414, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NAV3-20
Record Dates: First submitted 2016-08-02; First posted 2016-08-05 (Estimated); Last update posted 2017-03-15 (Actual); Status verified 2017-03

CONDITIONS: Anal Cancer
MeSH Terms: conditions — Anus Neoplasms | interventions — technetium-diethylenetriaminepentaacetic acid-mannosyl-dextran

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lymphoseek - 0.5 mCi, 50 ug (Experimental): A single dose of 50 µg Lymphoseek radiolabeled with 0.5 millicurie (mCi) (18.5 MBq) 99m Tc
  Interventions: Drug: Lymphoseek

INTERVENTIONS:
Drug: Lymphoseek

SUMMARY:
Prospective, open-label, within-subject, multi-center pilot study of Lymphoseek in the detection of lymph nodes in subjects with known squamous cell carcinoma of the anus.

DETAILED DESCRIPTION:
Prospective, open-label, within-subject, multi-center pilot study of Lymphoseek in the detection of lymph nodes in subjects with known squamous cell carcinoma of the anus. All subjects will receive a single dose of 50 µg Lymphoseek radiolabeled with 0.5 millicurie (mCi) (18.5 MBq) 99mTc.

ELIGIBILITY:
Inclusion Criteria:

* Subject has provided written informed consent with Health Insurance Portability and Accountability Act of 1996 (HIPAA) authorization
* Has histologically confirmed squamous cell carcinoma of the anus (anal canal or perianus)
* Has a documented clinical stage using the tumor, lymph node, metastasis staging (TNM) classification system that was established by at least physical exam with manual palpation, digital anorectal examination, high-resolution anoscopy and PET/CT imaging evaluation of the bilateral inguinal area
* Is at least 18 years of age at the time of consent
* Has an Eastern Cooperative Oncology Group (ECOG) performance status of Grade 0 to 3
* If of childbearing potential, the subject has a negative pregnancy test within 48 hours before administration of Lymphoseek, has been surgically sterilized, or has been postmenopausal for at least 1 year

Exclusion Criteria:

* The subject has had radiation therapy, chemotherapy or immunotherapy within the 30 days prior to Lymphoseek administration
* Has had previous surgery or node dissection (exclusive of fine needle aspiration) or radiation to node basins that would be involved in the intraoperative lymphatic mapping procedure
* Has a known allergy to dextran
* Is breast-feeding or pregnant
* Before the administration of Lymphoseek, has received any radiopharmaceutical within 7 radioactive half-lives of that radiopharmaceutical
* Has received an investigational product within the 30 days prior to Lymphoseek administration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-09; Primary Completion 2017-08 (Estimated); Study Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
Concordance (the proportion of the number of subjects with lymph nodes identified by Lymphoseek and standard of care methods compared to the number of subjects with lymph nodes identified by standard of care methods) | 2-5 Days

SECONDARY OUTCOMES:
Reverse Concordance (the proportion of the number of subjects with lymph nodes identified by Lymphoseek and standard of care methods compared to the number of subjects with lymph nodes identified by Lymphoseek) | 2-5 Days
Nodal Concordance (the proportion of the number lymph nodes identified by Lymphoseek and standard of care methods compared to the number of lymph nodes identified by standard of care methods) | 2-5 Days
Reverse Nodal Concordance (the proportion of the number lymph nodes identified by Lymphoseek and standard of care methods compared to the number of lymph nodes identified by Lymphoseek) | 2-5 Days
Incidence of Adverse Events | 5 Days

CONTACTS AND LOCATIONS:
Overall Officials: Michael Blue, MD, Study Director — Cardinal Health 414, LLC

IPD SHARING:
Plan to Share IPD: No